CLINICAL TRIAL: NCT02047799
Title: Effect of Vitamin D Supplementation on Blood Pressure in Elderly People
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidad de Colima (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SanchezC
Record Dates: First submitted 2014-01-26; First posted 2014-01-28 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: High Blood Pressure
Keywords: elderly people, high blood pressure, vitamin D.
MeSH Terms: conditions — Hypertension | interventions — Calcitriol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Calcitriol (Active Comparator): A daily dose of 1000 IU of cholecalciferol (administered as 1 capsule of 25 μg each)
  Interventions: Dietary Supplement: Calcitriol
- Control (Placebo Comparator): A daily dose of placebo (administered as 1 capsule )
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Calcitriol — Subjects whom were enrolled for 6 weeks of treatment with a daily dose of Calcitriol (1000 UI)
  Arms: Calcitriol
Dietary Supplement: Control — Subjects whom were enrolled for 6 weeks of treatment with a daily dose of Placebo
  Arms: Control

SUMMARY:
The prevalence and incidence of cardiovascular disease (such as Hypertension) increases exponentially with age (McDermott, 2007;) These diseases account for 30% of the global mortality (WHO, 2011). Vitamin D (VD) insufficiency affects as many as half of otherwise healthy adults in developed countries (Holick, 2007). VD is implicated in the control of blood pressure (BP) through inhibition of the renin-angiotensin system (Yamshchikov, 2009), although the role of VD supplementation for prevention and treatment of the HTA is controversial.The purpose of this study was to investigate if VD supplement in elderly people reduces the levels of BP.

DETAILED DESCRIPTION:
Study population Adults aged ≥ 60 years with essential hypertension were recruited through nursing homes and physical activity groups in the state of Colima, México. 45 subjects were assessed for eligibility at our out-patient clinic. We excluded subjects with impaired renal or hepatic function; also subjects who had been treated with vitamin D within the last three months.

None were on hormone replacement therapy, but we included subjects on anti-hypertensive for more than 10 years and the dosages were unchanged during the study. Before randomization, two subjects withdrew the informed consent because of personal reasons, and two subjects were excluded due to the diagnosis of severe hypertension.

Design The design was a double-blind, placebo controlled randomized clinical trial. The participants were randomly assigned using a computer-generated randomization code into two groups: group 1 (calcitriol group)with 22 subjects whom were enrolled for 6 weeks of treatment with a daily dose of 1000 IU of cholecalciferol (administered as 1 capsule of 25 μg each) and group 2 with 23 subjects (control group) whom received a similar placebo tablet for also 6 weeks.

During treatment, nine subjects (20%) left the trial due to personal reasons. All patients provided written informed consent. The study was conducted in accordance with the Declaration of Helsinki II and the guidance on Good Clinical Practice (GCP). Approval was obtained from the bioethics committee of the Faculty of Medicine from the University of Colima (FM014/2012).

Measurement At the screening visit prior to randomization, subjects had a routine clinical examination and data concerning medical history. BP was measured 3 consecutive days at the same time, using a kit integrated aneroid sphygmomanometer with stethoscope (medimetrics 5769) with the patient seated and with at least 5 min rest. The subjects with average BP >140/90 mm Hg were included in the study.

Once enrolled in the study groups, anthropometrics measurements were collected. The measurements performed were weight and height with light clothing and no shoes, and the indicator body mass index (kg/m2) was calculated. For the determination of serum 25(OH)D,two blood samples were collected in the morning after an overnight fast of minimum 8 h on the day of the randomization and at the end of the study.

The patients attended control visits every week for safety measures, adverse event registration and assessment of compliance.Returned pills were counted at each visit, and compliance was calculated as the percentage of used pills compared to the expected number.

Biochemistry Serum 25(OH)D concentration were measured with the use of competitive enzyme-linked immunosorbent assay (ELISA: immunodiagnostic, Bernheim, Germany) after solid-phase extraction (reference range: 17-53 pg/mL). The intra- and interassay CVs for the 2 Vitamin D metabolites were <7,0% and 9,0%, respectively.

Statistical Analysis The data were analyzed with the SPSS version 21. The variables studied were described as frequencies, percentages and as median (interquartile range); inferential statistics were performed with non parametric tests (Mann Whitney and related sample Wilcoxon test), and correlations between variables were analyzed by bivariate correlation analysis by Pearson's correlation. Statistical significance was set at a p value < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 60 years with essential hypertension.
* Subjects on anti-hypertensive for more than 10 years and the dosages were unchanged during the study.

Exclusion Criteria:

* Subjects who had been treated with vitamin D within the last three months.
* None were on hormone replacement therapy.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-04; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Difference of systolic and diastolic blood pressure | 6 weeks
  Difference between systolic and diastolic blood pressure before and after treatment.

SECONDARY OUTCOMES:
Difference of Serum 25-Hidroxyvitamin-D | 6 weeks
  Difference between 25-Hidroxyvitamin-D before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime A Bricio Barrios, Principal Investigator; Carmen A Sánchez Ramírez, MD, PhD, Study Director — Universidad de Colima; Alín J Palacios Fonseca, MS, Study Chair — Universidad de Colima; Mario del-Toro Equihua, PhD, Study Chair — Universidad de Colima
Locations (1):
- Facultad de Medicina-Universidad de Colima, Colima, Mexico

REFERENCES:
- [Background] McDermott MM. The international pandemic of chronic cardiovascular disease. JAMA. 2007 Mar 21;297(11):1253-5. doi: 10.1001/jama.297.11.1253. No abstract available. PMID 17374819
- [Background] WHO, World Heart Federation, World Stroke Organization. Global atlas on cardiovascular disease prevention and control. The Atlas of Heart Disease and Stroke. World Health Organization, 2011;8-13
- [Background] Holick MF, Smith E, Pincus S. Skin as the site of vitamin D synthesis and target tissue for 1,25-dihydroxyvitamin D3. Use of calcitriol (1,25-dihydroxyvitamin D3) for treatment of psoriasis. Arch Dermatol. 1987 Dec;123(12):1677-1683a. PMID 2825606
- [Background] Yamshchikov AV, Desai NS, Blumberg HM, Ziegler TR, Tangpricha V. Vitamin D for treatment and prevention of infectious diseases: a systematic review of randomized controlled trials. Endocr Pract. 2009 Jul-Aug;15(5):438-49. doi: 10.4158/EP09101.ORR. PMID 19491064
- [Derived] Bricio-Barrios JA Rd, Palacios-Fonseca AJ MSc, Del Toro-Equihua M, Sanchez-Ramirez CA. Effect of Calcitriol Supplementation on Blood Pressure in Older Adults. J Nutr Gerontol Geriatr. 2016 Oct-Dec;35(4):243-252. doi: 10.1080/21551197.2016.1206499. PMID 27897610